CLINICAL TRIAL: NCT03056235
Title: A Randomized, Within-subject, Placebo-controlled, Single-blind Study to Evaluate the Efficacy of ELAPR002f in Females and Males With Atrophic Acne Scars
Brief Title: A Study to Evaluate the Efficacy of ELAPR002f in Females and Males With Atrophic Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elastagen Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELAPR-P1D
Record Dates: First submitted 2017-02-09; First posted 2017-02-17 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Atrophic Acne Scar
Keywords: Atrophic acne scar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELAPR002f (Experimental): ELAPR002f is a tropoelastin gel cross-linked with derivatised hyaluronic acid
  Interventions: Device: ELAPR002f
- Saline control (Placebo Comparator): Saline
  Interventions: Device: Saline

INTERVENTIONS:
Device: ELAPR002f — 30mg/ml Tropoelastin cross-linked with derivatised hyaluronic acid
  Arms: ELAPR002f
Device: Saline — Saline control
  Arms: Saline control

SUMMARY:
The study is designed to evaluate the efficacy of two formulations of a cross-linked tropoelastin matrix given the product codes ELAPR002f (collectively referred to as ELAPR or ELAPR002) for the treatment of rolling atrophic acne scars when administered as intradermal implants.

DETAILED DESCRIPTION:
The study consists of a pre-screen visit followed by seven study visits. There will be a pre-screen visit where up to 30 potential study subjects will have 2D and 3D photographs taken of the candidate treatment fields to enable the Sponsor and Trial Centre staff to set practical guidelines for subject recruitment based on example atrophic acne scar images and published acne scar assessment scales. Subjects participating in the pre-screen period may be invited to participate in the full study if they are considered to be able to meet the eligibility criteria.

There will be a screening visit to confirm eligibility and to assess baseline parameters (D-28 to D-1). In addition, the proposed treatment fields on each side of the face will be selected at screening and recorded with 2D & 3D photographs and their location marked in detail on acetate sheets.

For enrolled subjects there will be three intradermal (i.d.) treatment sessions of ELAPR002f and placebo, given at one-monthly intervals (approximately D0, D28 and D56). The treatment at D0 will be administered so as to reduce the appearance of the atrophic rolling acne scars in the treatment field relative to the surrounding skin. The treatments at D28 and D56 will be given to optimise the treatment outcome and to minimise the appearance of the atrophic rolling acne scars in the treatment field.

In addition to the facial acne scars, a minimum of 5 subjects in each treatment group will also receive treatment on two moderate to severe, distensible, rolling acne scars present approximately 5-10cm apart on the back or torso.

There will be an assessment visit 14 and 84 days after the first treatment session (D14 and D84) to review any adverse events and assess the implant sites.

ELAPR002f will be administered alone vs. placebo. Subjects will be followed for a total of 24 weeks (to D168) following the first treatment, with efficacy and safety assessments undertaken at each study visit. At the final follow-up visit (D168) a biopsy sample will be taken from of each of the treated atrophic acne scars on the back or torso (active and placebo treated) from those subjects who received treatment to scars on the back or torso.

Each study subject will act as their own control with active and placebo treatments given single-blind to treatment fields on contralateral sides of the face. Prior to administration the selected treatment fields will be identified and marked with a washable marker using the 2D and 3D images and acetate sheets created at the screening visit to ensure consistency of anatomic sites for treatment (and biopsy for those subjects receiving treatment to the back or torso). Follow-up period extended to D336.

ELIGIBILITY:
Inclusion Criteria:

* Female/male subjects with matched treatment fields of approximately 2cm x 2cm on each side of the face on the temples or cheek bones that each contain a minimum of two rolling atrophic acne scars that are distensible when stretched between one's fingers and that are classified as moderate to severe on the scales detailed at Appendix 2.
* Acne scars in areas of otherwise normal healthy skin.
* Age: 18 - 55 years.
* Capable of providing voluntary informed consent.
* Good general health.
* Female subjects who are sexually active will be of non-child bearing potential (i.e., surgically sterilized or postmenopausal), abstain from sexual intercourse, or use a reliable method of contraception (e.g. hormonal contraceptive, condom, IUD) for at least 30 days prior to dosing and during the duration of the study.
* Fitzpatrick skin types I, II, III, IV or V.

Exclusion Criteria:

* No active ongoing acne lesions on the face (or back and torso for the subjects who will also receive treatment in these areas).
* Subjects who present with predominantly ice pick or box scars.
* Current or previous treatment of atrophic acne scars with fillers, lasers, or deep chemical peels which reach the dermis, or any other medical or surgical treatment which in the investigators opinion could reasonably be deemed to impact on the results of the current clinical study.
* Known hypersensitivity to tropoelastin, hyaluronic acid or any other component of ELAPR002f or ELAPR002g.
* Female subjects with a positive pregnancy test, women refusing to agree to adequate contraception and pregnancy tests during the study, or women who are planning to become pregnant during the period of the trial.
* Participation in a clinical trial of a pharmacological agent within 1 month prior to screening.
* Clinically significant haematology or biochemistry findings at screening.
* Positive test for hepatitis B, hepatitis C or HIV at screening.
* Bleeding diathesis, anticoagulant drugs, thrombocytopenia or clinically significant prolonged APTT or PT.
* Chronic use of aspirin, other non-steroidal anti-inflammatory drugs or other anti-platelet agents.
* History of keloid formation.
* History of granulomatous or connective tissue disease.
* Systemic corticosteroids within last 12 weeks.
* Currently using topical retinoids, or have used topical retinoids in the past 8 weeks.
* Diabetes or other metabolic disorders that may interfere with the subject's response to treatment in the opinion of the investigator.
* Any serious medical condition which in the opinion of the investigator would have a strong possibility of requiring systemic corticosteroid medication.
* Females who are pregnant or lactating.
* Previous administration of tropoelastin.
* A history of anaphylaxis or allergic reactions including any known hypersensitivity to lidocaine.
* Use of any investigational product on the intended implant site in the previous 12 months.
* Fitzpatrick skin types VI.
* Any other factor that in the opinion of the Investigator would make the subject unsafe or unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Measurement of the dimensions of acne scars pre and post treatment | 6 months
  The volume of acne scar depressions within the treatment field will be measured using 2D and 3D camera analysis

SECONDARY OUTCOMES:
Assessment of product integration into dermal tissue using histological analysis | 6 months
  Subjects who receive treatments to acne scars on the torso will undergo biopsy and the tissue analysed using histology techniques. Measure incidence and severity of implant site reactions as assessed by clinical observation and subject diary card records.

CONTACTS AND LOCATIONS:
Overall Officials: Frans Van den Berg, Doctor, Principal Investigator — Hammersmith Medical Research
Locations (1):
- Hammersmith Medicines Research, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No